CLINICAL TRIAL: NCT03037515
Title: A Randomized Controlled Trial of Oral and Intravenous Tranexamic Acid in Lumbar Spine Surgery
Brief Title: Oral and Intravenous Tranexamic Acid in Lumbar Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopaedic Spine Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10608
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Blood Loss, Surgical; Blood Loss Anemia
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous Tranexamic Acid (Active Comparator): The IV TXA group will receive the standard dosing for our institution of 1 g TXA (diluted in 100 mL normal saline) given as an IV bolus immediately before incision and another 1 g TXA given before closure.
  Interventions: Drug: Tranexamic Acid
- Oral Tranexamic Acid (Active Comparator): The oral TXA group will receive 1950 mg TXA (3 tablets of 650 mg) approximately 2 hours before incision.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — To identify if intravenous tranexamic acid is superior to oral tranexamic acid in reducing blood loss and need for transfusion in lumbar spine surgery.
  Other Names: Lysteda

SUMMARY:
The purpose of this project is to compare the effectiveness of two different but well accepted routes of administration of tranexamic acid in order to reduce blood loss and need for transfusion in patients undergoing lumbar spine surgery. Specifically, this study seeks to identify if intravenous tranexamic acid is superior to oral tranexamic acid in reducing blood loss and need for transfusion.

DETAILED DESCRIPTION:
Spine surgery is associated with large amount of perioperative blood loss. Factors influencing blood loss include surgical technique, operative time, number of vertebral levels arthrodesed, and others. Significant blood loss is associated with complications such as hypotension, end organ damage, or coagulopathy. Blood transfusions can increase risks of infection, blood incompatibility, and allergic reactions. Due to the significant risks and complications associated with blood loss and allogenic transfusions, efforts to identify safe and effective ways of lowering blood loss during spine surgery are crucial. Many methods have been utilized to reduce allogenic blood transfusions, such as autologous blood predonation, antifibrinolytic drugs, acute normovolemic hemodilution, intraoperative blood salvage, and others. Furthermore, the administration of antifibrinolytics, such as tranexamic acid (TXA) and epsilon-aminocaproic acid (EACA), has been shown to reduce bleeding in cardiac, gynecological, urologic and total joint replacement surgeries. There have been many published studies investigating various antifibrinolytic agents such as TXA, EACA, and aprotinin. While aprotinin was shown to increase mortality rate in patients following cardiac surgery, TXA and EACA have not been shown to cause any substantial morbidity or to increase rate of thromboembolic events. Although IV TXA has been shown to be effective in reducing blood loss and transfusions in patients undergoing spine surgery, no studies in the literature have investigated the efficacy of PO TXA in decreasing blood loss and transfusions. The investigators believe that PO TXA will be just as efficacious and more cost-effective in reducing blood loss and transfusion needs in patients undergoing lumbar spine surgery.

The ultimate goal is identifying the most cost-effective protocol to decrease blood loss and need for transfusion. If oral TXA is found to be as efficacious as IV TXA in reducing blood loss and need for transfusion, significant cost savings can be achieved for the patient and the health care system in general.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over age 18 and scheduled for open lumbar spine surgery (primary or revision)
* Must be able to swallow tablets

Exclusion Criteria

* Known allergy to TXA
* History of renal failure or kidney transplant
* History of arterial thromboembolic event (eg. myocardial infarction, stroke) within the past year
* Placement of an arterial stent within the past year
* History of blood clots (DVT, PE) within the past year
* Refusal to receive blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss between the two groups | Day of surgery to 1 day after surgery, up to 7 days
  For males: BV = 0.3669*(Height in meters)^3 + 0.03219*(Weight in kilograms) + 0.6041 For females: BV = 0.3561*(Height in meters)^3 + 0.03308*(Weight in kilograms) + 0.1833 Hbloss = BV*(Hbi-Hbe )*0.001 + Hbt Blood loss = 1000*(Hbloss/Hbi) Hbloss = Hemoglobin loss; BV = Blood Volume; Hbi = initial Hgb; Hbe = ending Hgb; Hbt = transfused Hgb = about 52g (SD 5.4g) per 1u pRBC (320mL)

SECONDARY OUTCOMES:
Post-operative drop in hemoglobin between the two groups | 1 day after surgery until patient is discharged, up to 7 days
Post-operative blood loss between the two groups | 1 day after surgery until patient is discharged, up to 7 days
Number of units transfused between the two groups | 1 day after surgery until patient is discharged, up to 7 days
Post-operative drain output between the two groups | 1 day after surgery until patient is discharged, up to 7 days
Incidence of thromboembolic events between the two groups | 1 day after surgery until patient returns for first postoperative visit (through study completion, an average of 4 weeks after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586